CLINICAL TRIAL: NCT06991452
Title: Multicenter Clinical Validation of a Novel Strategy for Early Diagnosis and Recurrence Monitoring in Colorectal Cancer
Brief Title: Early Diagnosis and Recurrence Monitoring of Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jie Liu, Professor, Huashan Hospital
Other Study IDs: KY2025-627
Record Dates: First submitted 2025-05-13; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Early diagnosis of colorectal cancer; Early warning of colorectal cancer recurrence; Liquid biopsy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Early colorectal cancer
  Interventions: Diagnostic Test: Liquid biopsy
- Control study participants with normal colonoscopy findings
  Interventions: Diagnostic Test: Liquid biopsy
- Patients with non-neoplastic intestinal diseases
  Interventions: Diagnostic Test: Liquid biopsy
- Patients with non-intestinal malignancies
  Interventions: Diagnostic Test: Liquid biopsy
- Colorectal cancer resistant to chemotherapy
  Interventions: Diagnostic Test: Liquid biopsy
- Patients with colorectal cancer liver metastasis
  Interventions: Diagnostic Test: Liquid biopsy
- Colorectal cancer liver metastasis cohort control group
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Serum protein profile, serum metabolic mass spectrometry, plasma cfDNA/cfRNA genomic and epigenomic assays, and serum tumor markers were performed. Patients were followed up for 3 years at a 3-month interval. Collect surgically removed colorectal cancer samples to construct PDX models if necessary.

SUMMARY:
Colorectal cancer (CRC) has an insidious onset and its survival rate is closely related to clinical stage. While the 5-year survival rate of stage I patients exceeds 90%, it drops to 14% in stage IV. In China, only 15.2% of CRC cases are diagnosed at stage I, far below the rate in developed countries like the United States (24.1%). Early detection and screening are key to reducing CRC mortality and improving patient outcomes. However, current screening methods-including colonoscopy, fecal immunochemical tests (FIT), and emerging stool or blood-based biomarkers-face limitations such as invasiveness, low sensitivity, high cost, or lack of large-scale clinical validation. Importantly, these methods fail to dynamically reflect tumor evolution or assess prognosis and treatment response.

Liquid biopsy has recently emerged as a promising non-invasive strategy for early cancer detection. It enables detection of tumor-related components in body fluids such as circulating tumor DNA (ctDNA), circulating tumor cells (CTCs), tumor-educated platelets (TEPs), exosomes, and cancer-specific proteins. These approaches offer a comprehensive view of tumor heterogeneity, epigenetic modifications, and treatment response. Our multidisciplinary team, from Fudan University, Xiamen University, and Xuzhou Medical University, has previously developed a cfDNA-5hmC-based diagnostic model using 5hmC-Seal technology, achieving 88% sensitivity and 89% specificity in detecting CRC.

To further improve tissue specificity and diagnostic accuracy, the investigators integrated multi-omics data and advanced AI techniques (including a Transformer-based deep learning model) to deconvolute tissue origin signals. In parallel, the investigators established a charge-selective CTC enrichment platform and discovered novel metabolic markers such as HPD that may indicate tumor recurrence and metastasis. The investigators team also developed a series of nano-biosensing platforms and tumor-targeting aptamer-based diagnostic kits, some of which have been granted national patents and clinical innovation awards.

This observational study will establish a large-scale, multi-center cohort of early-stage CRC patients. The investigators aim to construct a comprehensive multi-omics atlas from liquid biopsy samples, identify early diagnostic and prognostic biomarkers for CRC (including liver metastasis and drug resistance), and develop AI-driven models for non-invasive early detection and recurrence prediction. The study is expected to deliver clinically applicable technologies that improve CRC diagnostic accuracy, enable timely intervention, and reduce mortality. All study procedures will comply with ethical guidelines and be approved by institutional review boards.

ELIGIBILITY:
Inclusion Criteria:

1: Inclusion criteria for the case group:

1. Aged between 18 and 80 years old, regardless of gender.
2. Patients diagnosed with early colorectal cancer in our hospital, with the following specific criteria:

   1. Meet the diagnostic criteria of the Chinese Colorectal Cancer Diagnosis and Treatment Guidelines (2023 Edition) of the National Health Commission of the People's Republic of China, and be diagnosed with primary colorectal cancer by pathological tissue examination based on the imaging features of endoscopy, CT/CT enhanced scanning or MRI;
   2. Accept the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) Colorectal Cancer TNM Staging System (8th Edition, 2017) evaluation, and be evaluated as stage I or II colorectal cancer (T1-4N0M0).
   3. Have not received radiotherapy, chemotherapy, immunotherapy, surgery and other treatments.
3. No history of other malignant tumors.
4. Sign the informed consent form.

2: Inclusion criteria for participants in the control study with no obvious abnormalities in colonoscopy:

1. Aged between 18 and 80 years old, regardless of gender.
2. No abnormalities in colonoscopy results within the past 3 months.
3. No history of malignant tumors, no family history of malignant tumors (first-degree relatives, i.e. parents and/or second-degree relatives, i.e. grandfather, grandmother, uncle, etc., do not have malignant tumors).
4. No diseases such as obesity, hypertension, hyperlipidemia, metabolic syndrome, no bad living habits such as excessive drinking.
5. Voluntarily sign the informed consent form and can strictly follow the trial protocol to complete the study.

3: Inclusion criteria for patients with non-neoplastic intestinal diseases:

1. Aged between 18 and 80 years old, regardless of gender.
2. Patients diagnosed with non-neoplastic intestinal diseases such as colorectal adenoma and inflammatory bowel disease by colonoscopy and pathological examination. No history of colorectal cancer.

4: Inclusion criteria for patients with non-intestinal malignancies:

1. Aged between 18 and 80 years old, regardless of gender.
2. Meet the latest diagnostic criteria of the National Health Commission of the People's Republic of China or the Chinese Medical Association, and be diagnosed with non-intestinal malignancies such as gastric cancer, liver cancer, pancreatic cancer, esophageal cancer, etc. by pathological examination in our hospital based on imaging features of endoscopy, CT/CT enhanced scanning or MRI, combined with clinical manifestations and relevant laboratory tests. Have not received radiotherapy, chemotherapy, immunotherapy, surgery, etc. No history of colorectal cancer.

5: Inclusion criteria for the chemotherapy resistance prediction team:

1. Age between 18 and 80 years old, with no gender restrictions.
2. Patients diagnosed with colorectal cancer in our hospital, with specific criteria as follows:

   1. Meeting the diagnostic criteria of the "Diagnosis and Treatment Guidelines for Colorectal Cancer in China (2023 Edition)" issued by the National Health Commission of the People's Republic of China, and confirmed as primary colorectal cancer through pathological tissue examination based on endoscopic, CT/CT enhanced scan or MRI imaging features;
   2. Evaluated by the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) colorectal cancer TNM staging system (8th Edition, 2017), and assessed as stage II or III colorectal cancer (T1-4N1-2M0). c) Have not received radiotherapy, chemotherapy, immunotherapy, surgery or other treatments.
3. Evaluated as meeting surgical indications and planned to undergo radical surgery in three hospitals.
4. No history of other malignant tumors in the past.
5. Signed the informed consent form.

6: Inclusion Criteria for the Prediction Model of Colorectal Cancer Liver Metastasis:

1. Age between 18 and 80 years old, with no gender restrictions.
2. Patients diagnosed with colorectal cancer with liver metastasis in our hospital, with specific criteria as follows:

   1. Meeting the diagnostic criteria of the "Diagnosis and Treatment Guidelines for Colorectal Cancer in China (2023 Edition)" issued by the National Health Commission of the People's Republic of China, confirmed as primary colorectal cancer through endoscopy, liver ultrasound, CT/CT enhanced scan or MRI imaging features, and diagnosed with liver metastasis at the time of diagnosis;
   2. No previous treatment with radiotherapy, chemotherapy, immunotherapy, or surgery.
3. No history of other malignant tumors.
4. Signed informed consent form.

7: Inclusion criteria for the control group of the colorectal cancer liver metastasis cohort:

1. Age between 18 and 80 years old, with no gender restrictions.
2. Patients diagnosed with locally advanced colorectal cancer without distant metastasis in our hospital, with the following specific criteria:

   1. Meeting the diagnostic criteria of the "Diagnosis and Treatment Guidelines for Colorectal Cancer in China (2023 Edition)" issued by the National Health Commission of the People's Republic of China, and confirmed as primary colorectal cancer through pathological tissue examination based on endoscopic, CT/CT enhanced scan or MRI imaging features;
   2. Evaluated by the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) colorectal cancer TNM staging system (8th edition, 2017), the tumor invades the muscularis propria (T3), the perirectal fat (T4a), or adjacent organs (T4b), and/or has multiple local lymph node metastases (N1-2);
   3. Undergoing more than two imaging examinations (including liver ultrasound, enhanced CT, MRI, PET/CT, etc.), with no distant organ metastasis such as liver (M0) found; d) Have not received radiotherapy, chemotherapy, immunotherapy, surgery or other treatments.
3. No history of other malignant tumors in the past.
4. Signed informed consent.

Exclusion Criteria:

1. Severe complications, such as liver and kidney dysfunction (Child-Pugh C or eGFR<30).
2. Pregnant or lactating women.
3. Those who cannot accept venipuncture, are afraid of needles and blood, or have difficulty in blood collection.
4. Those who have donated blood (including blood products) or lost blood ≥200 mL in the past 2 months, or have received blood transfusions or used blood products in the past 2 months.
5. Those who have participated in any clinical trials of drugs or medical devices in the past 3 months or those whose trial drugs have not exceeded 5 half-lives (whichever is longer).
6. Unable to cooperate with follow-up (such as mental illness, expected survival <1 year).
7. Withdrawal or loss of follow-up during the study.
8. Incomplete information on study participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit a multi-center cohort of colorectal cancer patients (all stages), individuals with precancerous lesions (e.g., adenomas), and healthy controls. Participants must be ≥18 years old and capable of providing informed consent. This diverse population will enable training and external validation of a non-invasive AI-based diagnostic and prognostic model.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of a Novel Liquid Biopsy Model Incorporating Multi-Omics (Proteomics, Metabolomics, Circulating Nucleic Acid Analysis) and Serum Tumor Markers for Detecting Early-Stage Colorectal Cancer | November, 2027
Diagnostic Performance of Novel Liquid Biopsy Model Incorporating Multi-Omics (Proteomics, Metabolomics, Circulating Nucleic Acid Analysis) and Serum Tumor Markers for prediction of CRC recurrence | November, 2027
Diagnostic Performance of Novel Liquid Biopsy Model Incorporating Multi-Omics (Proteomics, Metabolomics, Circulating Nucleic Acid Analysis) and Serum Tumor Markers for prediction of CRC resistant to chemotherapy | November, 2027
Diagnostic Performance of Novel Liquid Biopsy Model Incorporating Multi-Omics (Proteomics, Metabolomics, Circulating Nucleic Acid Analysis) and Serum Tumor Markers for prediction of CRC metastasis. | November, 2027

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared but may be made available to qualified researchers upon reasonable request, subject to data use agreements and ethics approval, in accordance with participant consent and institutional policies.